CLINICAL TRIAL: NCT06419647
Title: Tracking Mood: The Effects of Daily Mood Tracking VAS on Alcohol Consumption in Adult Heavy Drinkers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ilona Myllyniemi (Other)
Collaborators: University of Cambridge (Other)
Responsible Party: Sponsor-Investigator, Ilona Myllyniemi, PhD Student, University of Cambridge
Organization: University of Cambridge (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MOODSTUDYALCOHOL
Record Dates: First submitted 2024-05-13; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Alcohol Abuse; Alcohol Drinking; Alcohol Use Disorder; Alcohol Dependence; Alcohol Intoxication
Keywords: Alcohol; AUD; Mood tracking; EMA; Emotional monitoring; Alcohol tracking
MeSH Terms: conditions — Alcoholism; Alcohol Drinking; Alcoholic Intoxication | interventions — Methods; Ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants complete daily mood tracking and weekly timeline followbacks of alcohol use
  Interventions: Behavioral: Intervention
- Control (No Intervention): Participants complete daily logs of time spent online and weekly timeline followbacks of alcohol use

INTERVENTIONS:
Behavioral: Intervention — Daily mood tracking tasks
  Other Names: Alcohol tracking; Mood tracking; Emotional monitoring; EMA
  Arms: Intervention

SUMMARY:
The study aims to investigate the effects that mood tracking may have on the alcohol consumption of adults who consume more than 20 UK units of alcohol per week, classifying as high-risk drinkers. The intervention group will track their mood on a daily basis with a visual analogue scale, while the control group will report their daily time spent online. The hypothesis, based on a series of prior pilot studies on alcohol tracking methods, is that mood tracking can reduce alcohol consumption in high-risk drinkers and therefore be a suitable addition to interventions related to decreasing alcohol consumption in heavy drinkers. The study will be conducted online through the Prolific platform.

DETAILED DESCRIPTION:
Participants will be recruited through Prolific. All participants will complete a series of demographic and psychometric questionnaires before beginning the study. Participants will also complete some of the psychometric questionnaires (RCQ, GAD-7, PHQ-9) at the end of the study to track any potential changes. Participants will be pre-screened for their motivation using a modified MTSS (Motivation to Stop Smoking) scale. Participants will also be asked to report their primary source of motivation regarding wanting to quit or reduce drinking, in addition to reporting their main goal regarding alcohol, where the options will be wanting to quit, wanting to reduce drinking, wanting to be more in control of their drinking, and not wanting to quit, reduce, or be more in control of drinking. All participants will also report their alcohol consumption using a timeline followback task with the ability to view both a calendar and a reference image of UK alcohol units. They'll report their alcohol consumption from the week before the study and complete two TLFBs during the study.

Intervention group participants complete daily visual analogue scales of their mood. Control group participants complete daily reports of how many hours they spent online the previous day.

ELIGIBILITY:
Inclusion Criteria:

* Speaking fluent English
* being over 18 years of age
* High completion rates of previous studies on the Prolific platform
* Being located in the United Kingdom
* Consuming over 20 UK units of alcohol per week

Exclusion Criteria:

* Having an ongoing mental health condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender options provided are as follows: Male, Female, Non-binary, Transgender man, Transgender woman, Other, Prefer not to say
Enrollment: 2000 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
TLFB | 3 weeks
  Timeline followbacks completed of consumed alcohol units reflecting alcohol units (UK) of alcohol consumed before the study and throughout the study

SECONDARY OUTCOMES:
GAD-7 | 3 weeks
  Comparison of potential changes in GAD-7 score before and after study
PHQ-9 | 3 weeks
  Comparison of potential changes in PHQ-9 score before and after study
RCQ | 3 weeks
  Comparison of potential changes in Readiness to Change score and Stage of Change destination before and after study

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Voon, PhD, MD, Study Director — University of Cambridge

IPD SHARING:
Plan to Share IPD: No
Study protocol, statistical analysis plan, informed consent form will be shared